CLINICAL TRIAL: NCT05062577
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of ASP8062 as an Add-on Therapy to Buprenorphine/Naloxone in Participants With Opioid Use Disorder
Brief Title: A Study to Assess the Safety and Efficacy of ASP8062 as an Add-on Therapy to Buprenorphine/Naloxone in Participants With Opioid Use Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to corporate strategic considerations
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8062-CL-2221
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
Keywords: ASP8062,; Opioid Use Disorder,; OUD,; Buprenorphine/Naloxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — ASP8062; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8062 in combination with buprenorphine/naloxone (Experimental): Participants will receive ASP8062 once daily at bedtime (QHS) and buprenorphine/naloxone once daily every morning (QAM) for 12 weeks.
  Interventions: Drug: ASP8062; Drug: buprenorphine/naloxone
- Placebo ASP8062 in combination with buprenorphine/naloxone (Placebo Comparator): Participants will receive matching placebo once daily at bedtime (QHS) and buprenorphine/naloxone once daily every morning (QAM) for 12 weeks.
  Interventions: Drug: Placebo ASP8062; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: ASP8062 — oral
  Arms: ASP8062 in combination with buprenorphine/naloxone
Drug: Placebo ASP8062 — oral
  Arms: Placebo ASP8062 in combination with buprenorphine/naloxone
Drug: buprenorphine/naloxone — sublingual

SUMMARY:
The purpose of this study is to evaluate the efficacy; safety and tolerability of ASP8062 compared with placebo ASP8062 as add-on therapy to buprenorphine/naloxone.

DETAILED DESCRIPTION:
The study will consist of the following periods: Screening Period (up to 56 days); Double-blind treatment period (12 weeks/ 85 days); a Buprenorphine/naloxone down-titration period (as determined by the participant in collaboration with the investigator) (14 days); and a Follow-up period (30 days post last dose ASP8062 or placebo ASP8062 for ASP8062 End of Treatment [EOT]).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of moderate or severe opioid use disorder (OUD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Ed (DSM-5) using the Mini International Neuropsychiatric Interview (MINI) version 7.02.
* Participant is voluntarily seeking treatment for OUD, and is either:

  * Currently receiving medication-assisted treatment (MAT) (buprenorphine/naloxone maintenance dose equivalent to 16 mg/4 mg sublingual for >=28 days prior to screening) for OUD and considered clinically unstable, defined as: currently misusing opioids and has at least 4 positive urine drug screens during the Screening Period (including morphine and metabolites, diacetylmorphine [heroin], codeine, oxycodone, hydrocodone, hydromorphone, fentanyl and metabolites, meperidine, propoxyphene, tramadol, oxymorphone and methadone)
  * Is not currently receiving MAT for OUD, and has not received MAT (consistently for > 48 hours) within 60 days prior to screening, and is: willing to initiate buprenorphine/naloxone therapy; considered to be a good candidate for buprenorphine/naloxone treatment based on medical and psychosocial history; able to tolerate buprenorphine/naloxone at the required maintenance dose of 16 mg/4 mg during the 7 days prior to randomization; has a positive urine drug screen at the initial screening visit (Visit 1) (including morphine and metabolites, diacetylmorphine (heroin), codeine, oxycodone, hydrocodone, hydromorphone, fentanyl and metabolites, meperidine, propoxyphene, tramadol, oxymorphone and methadone).
* Participant does not have on-going opioid withdrawal symptoms (a score of < 11 on the Clinical Opioid Withdrawal Scale (COWS)) at the time of randomization (Day 1).
* Participant has a body mass index range of 18.5 to 45.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Participant has stable living conditions.
* Participant agrees not to make significant changes to current non-medication therapy interventions (e.g., counseling, psychotherapy) in place at the time of Screening throughout the duration of the study.
* Participant agrees not to participate in another interventional study while participating in the present study; defined as from the time of informed consent form (ICF) signature until completion of the last study visit.
* Female participant is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational product (IP) administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female participant must not donate ova starting at screening and throughout the study period and for 30 days after final IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 90 days after final IP administration.
* Male participant must not donate sperm starting at screening and throughout the study period and for 90 days after final IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 90 days after final IP administration.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has a history of respiratory depression while on buprenorphine-based or other MAT for OUD.
* Participant has human immunodeficiency virus (HIV) per screening serology test.
* Participant has a positive hepatitis B surface antigen (HbsAg) or detectable hepatitis B DNA. Participants with negative HbsAg, positive hepatitis B core antibody (anti-HBc) and negative hepatitis B surface antibody (anti-HBs) are eligible if hepatitis B DNA is undetectable.
* Current diagnosis of chronic pain and currently treated with opioids other than buprenorphine or buprenorphine/naloxone.
* Current DSM-5 diagnosis of moderate to severe substance use disorder on any other psychoactive substances other than opioids, caffeine or nicotine (e.g., alcohol, sedatives) and the non-opioid substance use disorder(s) are considered primary or coprimary, causing current (last 30 days) significant impairment and/or would interfere with the efficacy and safety assessments.
* Participant has 2 or more positive urine drug screen (UDS) results for barbiturates or benzodiazepines during screening. (Day 1 eligibility will be based on a quick urine test conducted on-site, and not a sample sent to the central lab.)
* Participant has a known or suspected hypersensitivity to ASP8062, buprenorphine, naloxone or any components of the formulations used.
* Participant has previous exposure to ASP8062.
* Participant has a history of suicide attempt or suicidal behavior within 12 months prior to screening or has any suicidal ideation that meets criteria at a level of 4 or 5 by using the Columbia-Suicide Severity Rating Scale (C-SSRS) within 12 months prior to screening or who is at significant risk to commit suicide, as assessed at screening or at Day 1.
* Participant's prescription for buprenorphine/naloxone is unable to be filled at the pharmacy during Screening because they are already receiving an opioid based MAT.
* Participant has any clinically significant liver chemistry test result including aspartate aminotransferase [AST] or alanine aminotransferase [ALT] result > 3 times above the upper limit of normal (ULN), and total bilirubin [TBL] result > 1.5 times above the ULN at screening. These assessments may be repeated once, after a reasonable time period (but within the Screening Period).
* Participant has a mean pulse < 45 or > 110 beats per minute (unless above the upper bound of the range [> 110 beats per minute] deemed to be secondary to opioid withdrawal); resting systolic blood pressure > 140 mmHg or < 90 mmHg, and/or a resting diastolic blood pressure > 90 mmHg at screening (unless out of range blood pressure is deemed to be secondary to opioid withdrawal). These assessments may be repeated once after a reasonable time period (but within the Screening Period).
* Participant has a clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening or at randomization (Day 1). If the ECG is abnormal an additional ECG can be carried out. If this also gives a clinically significant abnormal result the participant must be excluded.
* Participant has a history of chest pain or palpitation with either exertion or drug use, myocardial infarction, endocarditis (within 12 months of screening), unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease or a family history of Long QT Syndrome.
* Participant has a clinically significant abnormality (e.g., severe respiratory insufficiency) in past medical history or at the screening visit that may place the participant at risk or interfere with the treatment outcomes.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) > 450 msec (for male participants) and > 470 msec (for female participants) at screening or at randomization. If the mean QTcF exceeds the limits above, one additional triplicate ECG can be taken on Day 1.
* Participant has known kidney disease and a glomerular filtration rate (GFR) < 60 mL/min per meter squared at screening.
* Participant has evidence of any clinically significant, uncontrolled cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary (including obstructive sleep apnea not controlled by a continuous positive airway pressure device), neurologic, dermatologic, psychiatric (other than moderate to severe OUD or other mild substance use disorders), renal and/or other major disease. Participants with mild, moderate or severe cocaine use disorder are not eligible.
* Participant has planned surgery during the study participation.
* Participant has an active malignancy or a history of malignancy (except for treated non melanoma skin cancer) within 5 years of screening.
* Participant's treatment for OUD was required by a court order, or participant's current incarceration or pending incarceration/legal action that could prohibit participation or compliance in the study.
* Participant is homeless or living in a shelter.
* Participant has manic-depressive illness or Major Depressive Disorder with psychotic features.
* Participant has clinically significant anemia or low hemoglobin (levels < 9 g/dL) at screening or donation of > 250 mL of blood or plasma within 30 days prior to providing informed consent.
* Participant is currently using protocol-specified prohibited medications and is unable to wash out or adjust their dosage.
* Participant has used any cytochrome P450 (CYP) 3A4 inhibitor (including most azole antifungals, macrolide antibiotics, protease inhibitors and antidepressants) or inducer (including phenobarbital, arbamazepine, phenytoin and rifampin) within 4 weeks prior to randomization.
* Participant has a negative lab test for buprenorphine and norbuprenorphine during screening (at any time prior to Day 1) for participants currently receiving treatment with buprenorphine/naloxone, or during the Run-in Period for participants newly initiating buprenorphine/naloxone treatment. The Day 1 collection will not be included in the eligibility assessment for either participant group.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant is an employee of the Astellas Group, the clinical research organization (CRO) involved or the investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child or sibling, whether biological or legally adopted).
* Participants with a positive urine drug screen for cocaine during Screening and/or a current diagnosis of mild, moderate or severe cocaine use disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with >= 80% of urine samples negative for misuse of opioid drugs combined with self-reports negative for opioid use | Up to 12 weeks
  Participants will undergo weekly assessments for misuse of opioid drugs through urine drug screening in combination with self-reports of opioid drug misuse.
  Percentage of participants with >= 80% of urine samples negative for misuse of opioid drugs combined with self reports negative for opioid use will be reported.
Number of participants with Adverse Events (AEs) | Up to 16 weeks
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study Investigational Product (IP) and other study treatments, whether or not considered related to the study IP and other study treatments. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study IP and other study treatments. This includes events related to the comparator and events related to the (study) procedures.
  An AE is considered "serious" if, the event: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important event.

SECONDARY OUTCOMES:
The cumulative distribution function (CDF) of the percentage of urine samples negative for misuse of opioid drugs combined with self-reports negative for opioid use | Up to 12 weeks
  Participants will undergo weekly assessments for misuse of opioid drugs through urine drug screening in combination with self-reports of opioid drug misuse.
  The cumulative distribution function (CDF) of the percentage of urine samples negative for misuse of opioid drugs combined with self-reports negative for opioid use will be reported.
Percentage of participants continuously abstinent from misuse of opioid drugs as assessed by urine samples and self-reports negative for opioid use | Up to 12 weeks
  Participants will undergo weekly assessments for misuse of opioid drugs through urine drug screening in combination with self-reports of opioid drug misuse.
  Percentage of participants continuously abstinent from misuse of opioid drugs as assessed by urine samples and self-reports negative for opioid use will be reported.
Total number of visits of abstinence from misuse of opioid drugs as assessed by urine samples and self-reports negative for opioid use | Up to 12 weeks
  Participants will undergo weekly assessments for misuse of opioid drugs through urine drug screening in combination with self-reports of opioid drug misuse.
  Total number of visits of abstinence from misuse of opioid drugs will be reported.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant vital sign values.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant laboratory values.
Change from baseline in blood oxygen saturation (SpO2) | Baseline and up to 16 weeks
  The blood oxygen saturation (SpO2) will be measured using a pulse oximeter placed on the participant's fingertip.
  Number of participants with low SpO2 levels will be reported.
Number of participants with Routine 12-lead electrocardiogram (ECG) abnormalities and/or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant Routine 12-lead ECG values.
Number of participants with suicidal ideation and/or suicidal behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 16 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior.
  Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported.
Overall mortality (including opioid overdose mortality) | Up to 16 weeks
  The number of participants for overall mortality and mortality due to opioid overdose will be summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.